CLINICAL TRIAL: NCT00500721
Title: An Open-Label, Single-Dose Desipramine, Multiple-Dose HCV-796, Sequential 3-Period Study to Determine the Pharmacokinetics of the Potential Drug Interaction Between HCV-796 and Desipramine
Brief Title: Study Evaluating the Pharmacokinetics of the Potential Drug Interaction Between HCV-796 and Desipramine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: ViroPharma (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 3173A1-1120
Record Dates: First submitted 2007-07-09; First posted 2007-07-13 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — HCV 796; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: HCV-796 — HCV-796 500mg BID x 14 days
Drug: Desipramine — Period 1: Single oral dose of desipramine (50 mg) on day 1. No test article administration on days 2 to 6.
  Period 2: Multiple oral doses of HCV-796 (500 mg) every 12 hours on days 1 to 9.
  Period 3: Multiple oral doses of HCV-796 (500 mg) every 12 hours on days 10 to 14 and a single oral dose of desipramine (50 mg) on day 10.

SUMMARY:
To evaluate the potential pharmacokinetic (PK) interaction of multiple oral doses of HCV-796 and a single dose of desipramine when coadministered to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) | 21 days

SECONDARY OUTCOMES:
Safety | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States